CLINICAL TRIAL: NCT01099228
Title: Combination Targeted Radiotherapy in Neuroendocrine Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Bushnell (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, David Bushnell, Professor, Radiology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200602763
Record Dates: First submitted 2010-03-26; First posted 2010-04-06 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine Tumor; Imaging
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 3-Iodobenzylguanidine; pentetreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 131-I MIBG and 111I-n pentetreotide (Active Comparator): 131-I MIBG and 111I-n pentetreotide
  Interventions: Other: 131-I MIBG and 111-In pentetreotide
- 131-I MIBG and In-111 DOTATATE (Active Comparator): 131-I MIBG and In-111 DOTATATE
  Interventions: Other: 131-I MIBG and In-111 DOTATATE

INTERVENTIONS:
Other: 131-I MIBG and 111-In pentetreotide — Subjects will receive 131I MIBG and 111In pentetreotide(surrogate for Y90-DOTATOC)
  Arms: 131-I MIBG and 111I-n pentetreotide
Other: 131-I MIBG and In-111 DOTATATE — 131I MIBG and In-111 DOTATATE (surrogate for 177Lu DOTATATE)
  Arms: 131-I MIBG and In-111 DOTATATE

SUMMARY:
The primary aim of this project is to determine, what fraction of individuals with neuroendocrine tumors would show substantially improved tumor dosimetry with combined agent therapy compared to "best" single agent therapy and determine the magnitude of the potential tumor radiation dose increase.

DETAILED DESCRIPTION:
RESEARCH PLAN / BACKGROUND AND SIGNIFICANCE:

Tumors originating from the neuroendocrine system, although relatively rare, may be life threatening. In cases where the disease has metastasized, the 5 year survival is very poor. 131I meta-iodobenzylguanidine (MIBG)and 90Y DOTA-D-Phe1-Tyr3-Octreotide (DOTATOC) are two radiopharmaceuticals that have shown promise as therapeutic agents in patients with metastatic neuroendocrine tumors. However, delivering sufficient radiation dose to the tumor to obtain objective anti-tumor responses or cure with these radiopharmaceuticals is challenging because of the allowable dose limits imposed by radiation damage to normal tissues. Organ biodistribution and kinetics of 90Y DOTATOC and 131I MIBG are substantially different, which leads to different critical organs for these agents, the kidney for Y90Y DOTATOC and the red marrow for 131I MIBG. We propose to investigate a mechanism to increase the radiation dose delivered to tumors without exceeding "critical" radiation dose to normal organs by combining 90Y DOTATOC and 131I MIBG.

AIMS / OBJECTIVES:

The primary aim of this project is to determine, what fraction of individuals with neuroendocrine tumors would show substantially improved tumor dosimetry with combined agent therapy compared to "best" single agent therapy and determine the magnitude of the potential tumor radiation dose increase.

METHODS:

To achieve this, we plan to perform serial scintigraphic imaging procedures to measure patient specific bone marrow, kidney, and tumor biodistribution and kinetics for 111In Pentetreotide and 131I-MIBG in adults and children with neuroendocrine tumors. Then, using the program we have already developed, we will input the individual dosimetry measures for bone marrow, kidney and tumor to determine the optimal amounts of administered radioactivity for the combination of 131I MIBG plus 90Y DOTATOC or 131I MIBG alone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with biopsy-proven metastatic (soft tissue) neuroendocrine tumors.
* Subjects with a Southwest Oncology Group (SWOG) performance score of 0-2 and an expected median survival of at least 6 months.
* The subject is able and willing to comply with study procedures and a signed and dated informed consent is obtained.
* Subjects must be >18 years of age

Exclusion Criteria:

* Subjects who use medications that are known to interfere with MIBG uptake and is unable to discontinue for medical reasons.
* Prior chemotherapy, radiotherapy or any investigational drugs within 60 days prior admission into this study. Patients must have recovered from all therapy-related toxicities
* Renal insufficiency with a serum creatinine 2 X ULN
* Subjects unable to lie still for the imaging studies.
* Subjects who because of their weight and body distribution do not fit into the imaging machine.
* Subjects receiving Sandostatin LAR < 21 days prior to dosing or Sandostatin Immediate Release (IR) < 24 hours prior to dosing.
* Female patients who are pregnant or breast feeding. Women of childbearing potential must have a negative serum/urine pregnancy test within 48 hours prior to administration of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Dosimetry Results | 1 week after scan
  Determine the patient specific bone marrow, kidney and tumor dosimetry results for each subject from the 2 groups will be used to calculate the optimal combination of administered activities for 131I-MIBG plus 90Y-DOTATOC (group 1) 131I-MIBG plus 177Lu-DOTATATE (group 2) and the resultant dose delivery to tumor from each combination

SECONDARY OUTCOMES:
Maximum Radiation Dose | 3 months
  Calculate the optimal amount for either agent when administered individually along with corresponding tumor radiation dose to determine the amount of each product will give maximum tumor kill and not damage other vunerable organs..

CONTACTS AND LOCATIONS:
Overall Officials: David Bushnell, M.D., Principal Investigator — University of Iowa; Veteran Affairs
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Department of Veteran Affairs Medical Center, Iowa City, Iowa